CLINICAL TRIAL: NCT06650332
Title: An Open-label, Multicohort Phase I/II Study of the Cadonilimab (AK104) Combination Regimen as First-line Treatment for HER2-expressing, Unresectable Locally Advanced or Metastatic Gastric (G) or Gastroesophageal Junction (GEJ) Cancer
Brief Title: Cadonilimab Combination Regimen as First-line Treatment for HER2-expressing GC/GEJ Patients
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Zhejiang Cancer Hospital (Other)
Responsible Party: Principal Investigator, Ying Jieer, Chief physician, Zhejiang Cancer Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AK104-IIT-C-M-0119
Record Dates: First submitted 2024-10-16; First posted 2024-10-21 (Actual); Last update posted 2024-10-21 (Actual); Status verified 2024-10

CONDITIONS: Metastatic HER2 Positive Gastroesophageal Junction Cancer
MeSH Terms: interventions — Trastuzumab; XELOX; disitamab vedotin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Cohort 1:AK104+trastuzumab+chemo (Experimental): AK104 (10 mg/kg, iv, Q3W, D1) in combination with trastuzumab (loading dose 8 mg/kg, iv, Q3W, D1; maintenance dose 6 mg/kg, iv, Q3W, D1) and chemotherapy (XELOX)
  Interventions: Drug: cadonilimab; Drug: Trastuzumab; Drug: XELOX
- Cohort 2:HER2-positive,AK104+RC48+chemo (Experimental): Phase Ⅰ:
  AK104:6mg/kg，iv，Q2W，D1 RC48:"3+3" design,1.5mg/kg、2.0mg/kg、2.5mg/kg chemotherapy:XELOX Phase Ⅱ:AK104 (6 mg/kg, iv, Q2W, D1) in combination with RC48 (recommended Phase I dose, iv, Q2W, D1) and chemotherapy (mFOLFOX6); PS:The chemotherapy treatment cycles will be determined by the investigator based on the participant's tolerability,and the maintenance treatment is AK104 in combination with RC48 and fluorouracil (5-FU) .
  Interventions: Drug: cadonilimab; Drug: Disitamab Vedotin; Drug: mFOLFOX6
- Cohort 3:HER2-expressing,AK104+RC48+chemo (Experimental): AK104:6mg/kg，iv，Q2W，D1 RC48:"3+3" design,1.5mg/kg、2.0mg/kg、2.5mg/kg chemotherapy:XELOX Phase Ⅱ:AK104 (6 mg/kg, iv, Q2W, D1) in combination with RC48 (recommended Phase I dose, iv, Q2W, D1) and chemotherapy (mFOLFOX6) PS:The chemotherapy treatment cycles will be determined by the investigator based on the participant's tolerability,and the maintenance treatment is AK104 in combination with RC48 and fluorouracil (5-FU) .
  Interventions: Drug: cadonilimab; Drug: Disitamab Vedotin; Drug: mFOLFOX6

INTERVENTIONS:
Drug: cadonilimab — Cohort 1:10 mg/kg, iv, Q3W, D1; Cohort 2/3:6 mg/kg, iv, Q2W, D1
  Other Names: AK104
Drug: Trastuzumab — loading dose 8 mg/kg, iv, Q3W, D1; maintenance dose 6 mg/kg, iv, Q3W, D1
  Arms: Cohort 1:AK104+trastuzumab+chemo
Drug: XELOX — Oxaliplatin: 130 mg/m\(^2\), IV, D1; Capecitabine: 1000 mg/m\(^2\), oral (PO), twice daily, D1-14.
  Arms: Cohort 1:AK104+trastuzumab+chemo
Drug: Disitamab Vedotin — 1.5、2.0、2.5mg/kg，IV，D1，Q2W
  Other Names: RC48
  Arms: Cohort 2:HER2-positive,AK104+RC48+chemo; Cohort 3:HER2-expressing,AK104+RC48+chemo
Drug: mFOLFOX6 — Oxaliplatin 85 mg/m\(^2\), IV, d1; Leucovorin (folinic acid) 400 mg/m\(^2\), IV, d1; 5-FU 400 mg/m\(^2\), IV, d1, followed by 2400 mg/m\(^2\), continuous intravenous infusion over 46 hours.
  Arms: Cohort 2:HER2-positive,AK104+RC48+chemo; Cohort 3:HER2-expressing,AK104+RC48+chemo

SUMMARY:
This trial is An open-label, multicohort, multicenter clinical study aimed at evaluating the efficacy and safety of the cadonilimab combination regimen in the treatment of advanced HER-2 positive gastric/gastroesophageal junction tumors

DETAILED DESCRIPTION:
This is a phase Ⅰ/Ⅱ clinicaltrial. Phase I aims to determine the maximum tolerated dose (MTD) or, if the MTD is not reached, the maximum administered dose (MAD) of AK104 in combination with RC48 (disitamab vedotin) as first-line treatment for unresectable locally advanced or metastatic GC/GEJ cancer, as well as the recommended phase II dose (RP2D).

Phase II aims to evaluate the efficacy and safety of AK104 in combination with trastuzumab and chemotherapy as first-line treatment for HER2-positive, unresectable locally advanced or metastatic GC/GEJ cancer; as well as the efficacy and safety of AK104 in combination with RC48 (disitamab vedotin) and chemotherapy as first-line treatment for HER2-expressing, unresectable locally advanced or metastatic GC/GEJ cancer.

ELIGIBILITY:
Inclusion Criteria:

-

1.Sign the informed consent form. 2. ≥18 years and ≤75 years . 3.Histologically confirmed unresectable locally advanced or metastatic gastric or gastroesophageal junction adenocarcinoma (tumor center located within 5 cm proximally or distally from the esophagogastric junction according to the Siewert classification system).

4.Confirmed PD-L1 expression status (accepts PD-L1 expression test results confirmed by the investigator).

5.HER2 expression (accepts HER2 expression test results confirmed by the investigator):

* Cohort 1 and Cohort 2: HER2-positive defined as IHC 3+, or IHC 2+ and ISH or FISH positive. ISH positivity is defined as a HER2 gene copy number to CEP17 copy number ratio ≥2.0; if the ratio is <2.0 but the HER2 gene copy number >6, it is also considered ISH positive.
* Cohort 3: HER2 low expression, defined as IHC 1+ or IHC 2+ but ISH or FISH negative.

  6.No prior systemic anti-tumor therapy. 7.With at least one measurable lesion (RECIST 1.1 criteria) in the subject . 8.Expected survival ≥ 3 months. 9.ECOG 0/1. 10.Adequate organ function is determined by the following criteria:
  1. Hematological (no transfusions or growth factor support allowed within 7 days before the first dose):Absolute neutrophil count (ANC) ≥ 1.5 × 10^9/L (1,500/mm³); Platelet count ≥ 100 × 10^9/L (100,000/mm³);Hemoglobin ≥ 90 g/L or ≥ 5.6 mmol/L.
  2. Liver:Serum albumin ≥ 28 g/L (no albumin infusions allowed within 14 days before the first dose);Total bilirubin (TBil) ≤ 1.5 × ULN; for subjects with liver metastases or evidence/suspicion of Gilbert's disease, TBil ≤ 3 × ULN; Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 2.5 × ULN; for subjects with liver metastases, AST and ALT ≤ 5 × ULN.
  3. Renal:Serum creatinine ≤ 1.5 × ULN or calculated creatinine clearance (CrCl) ≥ 50 mL/min (calculated using the Cockcroft-Gault formula);Urinalysis: urine protein < 2+; if urine protein ≥ 2+, then 24-hour urine protein ≤ 1 g.
  4. Coagulation:International normalized ratio (INR) ≤ 1.5 × ULNActivated partial thromboplastin time (aPTT) ≤ 1.5 × ULN;Prothrombin time (PT) ≤ 1.5 × ULN.
  5. Cardiac function:New York Heart Association (NYHA) class < III;Left ventricular ejection fraction (LVEF) ≥ 50%.

  11.For premenopausal women, a negative serum pregnancy test must be confirmed within 7 days before the first dose, and they must agree to use effective contraception during the study drug administration period and for 120 days after the last dose.

  12.Compliance with the trial schedule and follow-up procedures

Exclusion Criteria:

1. Known squamous cell carcinoma, undifferentiated carcinoma, or other histological types of gastric cancer, or adenocarcinoma mixed with other histological types.
2. Patients with gastric cancer without HER2 expression.
3. Known active or untreated brain metastases, leptomeningeal metastases, spinal cord compression, or leptomeningeal disease.
4. History of gastrointestinal perforation or fistula within 6 months before the first dose. Eligible if the perforation or fistula has been surgically repaired and the investigator judges the condition to be resolved or stable.
5. Active diverticulitis, abdominal abscess, or gastrointestinal obstruction.
6. Inability to swallow, malabsorption syndrome, or uncontrolled nausea, vomiting, diarrhea, or other significant gastrointestinal conditions that affect drug intake and absorption.
7. Clinically significant bleeding events or clear predisposition to bleeding within 1 month before the first dose, such as gastrointestinal bleeding, bleeding gastric ulcers (with active bleeding signs on endoscopy), or vasculitis.
8. Symptomatic moderate to severe ascites requiring therapeutic paracentesis (exceptions include asymptomatic ascites detected only on imaging). Uncontrolled or moderate to large pleural effusions, pericardial effusions.
9. Signs or symptoms of unacceptable worsening of primary disease during screening, as judged by the investigator.

   Exclusion Criteria due to Concurrent Diseases or Comorbid Conditions:
10. Active or documented history of inflammatory bowel disease (such as Crohn's disease or ulcerative colitis).
11. Major surgery within 4 weeks before the start of study treatment that has not fully recovered, or anticipated need for major surgery during the study period.
12. Uncontrolled systemic diseases, including but not limited to diabetes, hypertension, pulmonary fibrosis, acute lung disease, interstitial lung disease, decompensated cirrhosis, nephrotic syndrome, angina pectoris, severe arrhythmias, uncontrolled metabolic disorders, severe active peptic ulcer disease or gastritis.
13. Diagnosis of any malignancy other than gastric cancer within 5 years prior to entering the study.
14. Severe neurological or psychiatric disorders, including dementia, depression, and epilepsy.
15. Pregnant or breastfeeding women or individuals planning to conceive.
16. Presence of cardiovascular disease or cardiovascular risk factors.

    Drug Treatment-Related Exclusion Criteria:
17. Palliative radiotherapy for non-target lesions for symptom control is permitted, provided it was completed at least 2 weeks before the start of study treatment and any radiotherapy-induced adverse events have not resolved to ≤CTCAE Grade 1.
18. Prior treatment with immune checkpoint inhibitors, immune checkpoint agonists, immune cell therapies, or any other antibody-drug conjugates targeting tumor immune mechanisms.
19. Palliative local treatment for non-target lesions or systemic nonspecific immunomodulatory treatments (e.g., interleukins, interferons, thymosin) or traditional Chinese medicine/herbal remedies with antitumor indications within 2 weeks before the first dose.
20. Toxicities from prior anticancer therapy have not resolved to ≤CTCAE Grade 1, except for:

    1. Alopecia.
    2. Pigmentation changes.
    3. Peripheral neuropathy that has resolved to <CTCAE Grade 2.
    4. Late effects of radiotherapy that are unlikely to resolve, as judged by the investigator.
21. Requires systemic treatment with corticosteroids (>10 mg/day prednisone or equivalent) or other immunosuppressive drugs within 14 days before the first dose, except for:

    1. Inhalational, ophthalmic, topical corticosteroids or ≤10 mg/day prednisone or equivalent if no active autoimmune disease.
    2. Physiologic doses of systemic corticosteroids ≤10 mg/day prednisone or equivalent.
    3. Corticosteroids as premedication for infusion-related or allergic reactions (e.g., before CT scans).
22. Known history of severe hypersensitivity reactions to other monoclonal antibodies or known allergy or hypersensitivity to any of the study drugs or their components.
23. Known contraindications to oxaliplatin and capecitabine (Cohort 1); known contraindications to oxaliplatin, fluorouracil, and leucovorin (Cohorts 2 and 3).

    Exclusion Criteria for Special Immunological Status or Infections:
24. Active autoimmune disease requiring systemic therapy within 2 years before the start of study treatment, or an autoimmune disease that the investigator judges may recur or require treatment.
25. Known interstitial lung disease or non-infectious pneumonia that is currently symptomatic or required systemic corticosteroid treatment in the past, or that the investigator judges may impact the assessment or management of treatment-related toxicities.
26. Active infection, including infections requiring intravenous antibiotics or antifungal therapy within 2 weeks before dosing, fever of unknown cause during screening (CTCAE ≥ Grade 1, excluding fever due to tumor as judged by the investigator).
27. Subjects who are planned for or have undergone solid organ transplantation or allogeneic hematopoietic stem cell transplantation.
28. Active hepatitis B or active hepatitis C.
29. Known history of immunodeficiency or positive HIV test result.
30. Receipt of live vaccine within 28 days before the first dose, or plans to receive a live vaccine during the study.

    Other Exclusion Criteria:
31. Currently participating in another clinical study, unless it is observational, non-interventional, or in the follow-up phase of an interventional study.
32. Any condition that, in the investigator's judgment, may increase the risk of receiving the study drug or interfere with the evaluation of the study drug, the safety of the participant, or the interpretation of study results.
33. Participants who are not compliant with the requirements of this clinical trial or who have other factors that make them unsuitable for participation, as judged by the investigator.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2024-07-10 (Actual); Primary Completion 2026-08-10 (Estimated); Study Completion 2027-12-30 (Estimated)

PRIMARY OUTCOMES:
DLT | 28 days after the first dose
  Within 28 days after the first dose, adverse reactions related to Vicinium, including Grade 4 or higher hematologic toxicities or Grade 3 or higher non-hematologic toxicities (excluding alopecia), as graded by NCI CTCAE v5.0
Objective response rate(ORR) | up to 12 months
  The number of cases in which tumor size is reduced to PR or CR / the total number of evaluable cases (%)

SECONDARY OUTCOMES:
Progression-free survival (PFS) | up to 24 months
  Refers to the date from the date of admission to the date of the first progression of disease or death of any cause, using Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST v1.1).
Disease control rate (DCR) | up to 12 months
  Percentage of confirmed cases including complete remission (CR), partial remission (PR) and disease stability (SD) among patients with evaluable efficacy
Overall survival (OS) | up to 3 years
  The time interval between the start date of study drug and the date of death (any cause)
Adverse Events | [up to 24 months after enrollment or study close]
  Number and percentage of participants with Adverse Events(any grade)

CONTACTS AND LOCATIONS:
Overall Officials: Jieer Ying, MD, Principal Investigator — Zhejiang Cancer Hospital
Locations (1):
- Zhejiang Cancer Hospital, Hangzhou, Zhejiang, China